CLINICAL TRIAL: NCT06449092
Title: The Significance of Remnant Cholesterol and Carotid Intima Media Thickness in Patients With MAFLD
Acronym: MAFLD
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Khaled Mohammed, Ahmed Khaled Mohammed, Assiut University
Other Study IDs: Severity of MAFLD
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Detect the Significance of Remnant Cholesterol in Detection Severity of MAFLD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lipid profile — carotid intima media thickness
  Other Names: color doppler

SUMMARY:
1. To detect the significance of remenant cholesterol in detection severity of MAFLD
2. To detect the significance of carotid intima-media thickness in MAFLD

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is fatty infiltration of the liver in the absence of other causes of steatosis, such as alcohol consumption characterized by excessive fat accumulation in liver >5-10% of its weight encompassing a spectrum of increasingly severe clinico-pathological conditions - nonalcoholic fatty liver (NAFL) and nonalcoholic steato-hepatitis (NASH) with or without fibrosis/cirrhosis. Since NAFLD is frequently associated with further metabolic comorbidities such as obesity, type 2 diabetes mellitus, or dyslipidemia, it is generally considered as the hepatic manifestation of the metabolic syndrome A growing body of evidence also indicates that NAFLD is strongly associated with an increased risk of major CVD events and other cardiac complications (ie, cardiomyopathy, cardiac valvular calcification and cardiac arrhythmias), independently of traditional cardiovascular risk factors NAFLD has also been associated with an increase in the carotid intima- media thickness (CIMT), independent of conventional CVD risk factors. CIMT is a marker of early atherosclerosis and has been shown to predict increased risks of myocardial in-farction and stroke Fatty liver index (FLI) has been proposed as an accurate, convenient, and economic surrogate of the severity of NAFLD. Remnant cholesterol refers to the cholesterol content carried by triglyceride-rich lipoproteins, which include non-LDL-C and nonhigh density lipoprotein-cholesterol (HDL-C) A large number of studies have reported that serum remnant cholesterol levels were positively associated with the risk of coronary artery disease NAFLD

, type 2 diabetes , and metabolic syndrome

ELIGIBILITY:
Inclusion Criteria:

* The study will include adult patients (≥18 years) presented to fibroscan clinic and diagnosed as MAFLD.

Exclusion Criteria:

1. Patients Known previous cardiac disease ( cardiovascular disease, heart failure, arrhythmia )
2. Patients Known liver cirrhosis
3. septic patients
4. Patients have malignancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include patients presented to Fibroscan clinic, Internal medicine department at Assiut University hospitals within 1 year
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
To detect the significance of remnant cholesterol in detection severity of MAFLD | From Jan 2025 to Jan 2026
  lipid profile in MAFLD patients to detect remnant cholesterol
To detect the relationship between carotid intima-media thickness and remnant cholesterol in MAFLD and prediction of cardiovascular effect. | From Jan 2025 to Jan 2026
  color doppler and echocardiography in MAFLD patients

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided